CLINICAL TRIAL: NCT01439880
Title: A Multicenter, Controlled, Open-label Extension (OLE) Study to Assess the Long-term Safety and Efficacy of AMG 145 (Evolocumab)
Brief Title: Open Label Study of Long Term Evaluation Against LDL-C Trial
Acronym: OSLER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20110110; 2011-001915-29 (EudraCT Number)
Record Dates: First submitted 2011-09-22; First posted 2011-09-23 (Estimated); Results first posted 2019-07-10 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Hypercholesterolemia
Keywords: High cholesterol; Raised cholesterol; Cholesterol; Elevated Cholesterol
MeSH Terms: conditions — Hypercholesterolemia | interventions — evolocumab; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care (Active Comparator): Participants received standard of care (SOC) treatment for the first year of the study (SOC-controlled period). At week 52 participants began treatment with evolocumab 420 mg once a month (QM) for 4 years during the all-investigational product [all-IP] period.
  Interventions: Biological: Evolocumab; Other: Standard of care
- Evolocumab + SOC (Experimental): Participants received evolocumab 420 mg once a month plus standard of care for the first year of the study (SOC-controlled period). At week 52 participants continued treatment with evolocumab 420 mg QM for another 4 years during the all-IP period.
  Interventions: Biological: Evolocumab

INTERVENTIONS:
Biological: Evolocumab — Administered by subcutaneous injection
  Other Names: AMG 145; Repatha
Other: Standard of care — Standard of care therapy as per local practices. This could include prescribed therapies and/or dietary/exercise regimes
  Arms: Standard of Care

SUMMARY:
The primary clinical hypothesis is that long-term exposure of evolocumab (AMG 145) will be safe and well tolerated in adults with hypercholesterolemia.

ELIGIBILITY:
Inclusion Criteria:

* Complete a qualifying evolocumab (AMG 145) parent study protocol, including: 20101154 (NCT01375777), 20101155 (NCT01380730), 20090158 (NCT01375751), 20090159 (NCT01375764), and 20110231 (NCT01652703)

Exclusion Criteria:

* Experienced a treatment-related serious adverse event that led to investigational product (IP) discontinuation in the parent study
* Have an unstable medical condition, in the judgment of the investigator
* Known sensitivity to any of the products to be administered during dosing
* Currently enrolled in another investigational device or drug study (excluding evolocumab (AMG 145) parent study), or less than 30 days since ending another investigational device or drug study(s),or receiving other investigational agent(s)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1324 (Actual)
Dates: Start 2011-10-07 (Actual); Primary Completion 2018-06-20 (Actual); Study Completion 2018-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (167):
- United States (69):
  - Research Site, Birmingham, Alabama
  - Research Site, Tucson, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Malvern, Arkansas
  - Research Site, Anaheim, California
  - Research Site, Carmichael, California
  - Research Site, Inglewood, California
  - Research Site, Mission Viejo, California
  - Research Site, Newport Beach, California
  - Research Site, Thousand Oaks, California
  - Research Site, Tustin, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Littleton, Colorado
  - Research Site, Daytona Beach, Florida
  - Research Site, DeLand, Florida
  - Research Site, Green Cove Springs, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Melbourne, Florida
  - Research Site, Miami, Florida
  - Research Site, Ponte Vedra, Florida
  - Research Site, Port Charlotte, Florida
  - Research Site, Sanford, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Savannah, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Munster, Indiana
  - Research Site, Iowa City, Iowa
  - Research Site, Louisville, Kentucky
  - Research Site, Auburn, Maine
  - Research Site, Portland, Maine
  - Research Site, Bethesda, Maryland
  - Research Site, Chevy Chase, Maryland
  - Research Site, Brockton, Massachusetts
  - Research Site, Marquette, Michigan
  - Research Site, Brooklyn Center, Minnesota
  - Research Site, Tupelo, Mississippi
  - Research Site, Great Falls, Montana
  - Research Site, Henderson, Nevada
  - Research Site, Las Vegas, Nevada
  - Research Site, Cortlandt Manor, New York
  - Research Site, Endwell, New York
  - Research Site, New York, New York
  - Research Site, Williamsville, New York
  - Research Site, Raleigh, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Fargo, North Dakota
  - Research Site, Akron, Ohio
  - Research Site, Cadiz, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Norman, Oklahoma
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Camp Hill, Pennsylvania
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, York, Pennsylvania
  - Research Site, Mt. Pleasant, South Carolina
  - Research Site, Rapid City, South Dakota
  - Research Site, Bristol, Tennessee
  - Research Site, Arlington, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Norfolk, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Renton, Washington
  - Research Site, Seattle, Washington
  - Research Site, Tacoma, Washington
- Australia (4):
  - Research Site, Camperdown, New South Wales
  - Research Site, Maroubra, New South Wales
  - Research Site, Sydney, New South Wales
  - Research Site, Perth, Western Australia
- Belgium (8):
  - Research Site, Anthée
  - Research Site, Brussels
  - Research Site, Gozée
  - Research Site, Gribomont
  - Research Site, Halen
  - Research Site, Ham
  - Research Site, Linkebeek
  - Research Site, Uccle
- Canada (17):
  - Research Site, Kelowna, British Columbia
  - Research Site, Bay Roberts, Newfoundland and Labrador
  - Research Site, Mount Pearl, Newfoundland and Labrador
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Cambridge, Ontario
  - Research Site, Greater Sudbury, Ontario
  - Research Site, London, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, Sarnia, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Woodstock, Ontario
  - Research Site, Chicoutimi, Quebec
  - Research Site, Gatineau, Quebec
  - Research Site, Granby, Quebec
  - Research Site, Lachine, Quebec
  - Research Site, Pointe-Claire, Quebec
  - Research Site, Québec, Quebec
- Czechia (7):
  - Research Site, Brno
  - Research Site, Olomouc
  - Research Site, Prague
  - Research Site, Slaný
  - Research Site, Svitavy
  - Research Site, Ústí nad Orlicí
  - Research Site, Znojmo
- Denmark (3):
  - Research Site, Aalborg
  - Research Site, Ballerup Municipality
  - Research Site, Vejle
- Finland (2):
  - Research Site, Helsinki
  - Research Site, OYS
- Germany (2):
  - Research Site, Berlin
  - Research Site, Cologne
- Research Site, New Territories, Hong Kong
- Hungary (8):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Dunaújváros
  - Research Site, Gyula
  - Research Site, Kecskemét
  - Research Site, Komárom
  - Research Site, Szolnok
  - Research Site, Zalaegerszeg
- Japan (28):
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Fukui-shi, Fukui
  - Research Site, Kasuga-shi, Fukuoka
  - Research Site, Fujioka-shi, Gunma
  - Research Site, Maebashi, Gunma
  - Research Site, Takasaki-shi, Gunma
  - Research Site, Kawanishi-shi, Hyōgo
  - Research Site, Kobe, Hyōgo
  - Research Site, Hitachi-shi, Ibaraki
  - Research Site, Koga-shi, Ibaraki
  - Research Site, Mito, Ibaraki
  - Research Site, Komatsu-shi, Ishikawa-ken
  - Research Site, Takamatsu, Kagawa-ken
  - Research Site, Kochi, Kochi
  - Research Site, Kyoto, Kyoto
  - Research Site, Ina-shi, Nagano
  - Research Site, Matsumoto-shi, Nagano
  - Research Site, Suwa-shi, Nagano
  - Research Site, Ibaraki-shi, Osaka
  - Research Site, Toyonaka-shi, Osaka
  - Research Site, Hanyu-shi, Saitama
  - Research Site, Sayama-shi, Saitama
  - Research Site, Toda-shi, Saitama
  - Research Site, Chiyoda-ku, Tokyo
  - Research Site, Hachioji-shi, Tokyo
  - Research Site, Itabashi-ku, Tokyo
  - Research Site, Shinagawa-ku, Tokyo
  - Research Site, Toshima-ku, Tokyo
- Netherlands (3):
  - Research Site, Amsterdam
  - Research Site, Hoorn
  - Research Site, Utrecht
- Research Site, Oslo, Norway
- Research Site, Singapore, Singapore
- South Africa (4):
  - Research Site, Johannesburg, Gauteng
  - Research Site, Midrand, Gauteng
  - Research Site, Observatory, Western Cape
  - Research Site, Parow, Western Cape
- Spain (5):
  - Research Site, Córdoba, Andalusia
  - Research Site, Zaragoza, Aragon
  - Research Site, Barcelona, Catalonia
  - Research Site, Reus, Catalonia
  - Research Site, Madrid
- Sweden (3):
  - Research Site, Gothenburg
  - Research Site, Lund
  - Research Site, Stockholm
- Research Site, London, United Kingdom

REFERENCES:
- [Background] Koren MJ, Sabatine MS, Giugliano RP, Langslet G, Wiviott SD, Kassahun H, Ruzza A, Ma Y, Somaratne R, Raal FJ. Long-term Low-Density Lipoprotein Cholesterol-Lowering Efficacy, Persistence, and Safety of Evolocumab in Treatment of Hypercholesterolemia: Results Up to 4 Years From the Open-Label OSLER-1 Extension Study. JAMA Cardiol. 2017 Jun 1;2(6):598-607. doi: 10.1001/jamacardio.2017.0747. PMID 28291870
- [Background] Koren MJ, Giugliano RP, Raal FJ, Sullivan D, Bolognese M, Langslet G, Civeira F, Somaratne R, Nelson P, Liu T, Scott R, Wasserman SM, Sabatine MS; OSLER Investigators. Efficacy and safety of longer-term administration of evolocumab (AMG 145) in patients with hypercholesterolemia: 52-week results from the Open-Label Study of Long-Term Evaluation Against LDL-C (OSLER) randomized trial. Circulation. 2014 Jan 14;129(2):234-43. doi: 10.1161/CIRCULATIONAHA.113.007012. Epub 2013 Nov 19. PMID 24255061
- [Background] Daviglus ML, Ferdinand KC, Lopez JAG, Wu Y, Monsalvo ML, Rodriguez CJ. Effects of Evolocumab on Low-Density Lipoprotein Cholesterol, Non-High Density Lipoprotein Cholesterol, Apolipoprotein B, and Lipoprotein(a) by Race and Ethnicity: A Meta-Analysis of Individual Participant Data From Double-Blind and Open-Label Extension Studies. J Am Heart Assoc. 2021 Jan 5;10(1):e016839. doi: 10.1161/JAHA.120.016839. Epub 2020 Dec 16. PMID 33325247
- [Background] Hovingh GK, Raal FJ, Dent R, Stefanutti C, Descamps O, Masana L, Lira A, Bridges I, Coll B, Sullivan D. Long-term safety, tolerability, and efficacy of evolocumab in patients with heterozygous familial hypercholesterolemia. J Clin Lipidol. 2017 Nov-Dec;11(6):1448-1457. doi: 10.1016/j.jacl.2017.09.003. Epub 2017 Sep 22. PMID 29066265
- [Background] Koren MJ, Sabatine MS, Giugliano RP, Langslet G, Wiviott SD, Ruzza A, Ma Y, Hamer AW, Wasserman SM, Raal FJ. Long-Term Efficacy and Safety of Evolocumab in Patients With Hypercholesterolemia. J Am Coll Cardiol. 2019 Oct 29;74(17):2132-2146. doi: 10.1016/j.jacc.2019.08.1024. PMID 31648705
- [Background] Kasichayanula S, Grover A, Emery MG, Gibbs MA, Somaratne R, Wasserman SM, Gibbs JP. Clinical Pharmacokinetics and Pharmacodynamics of Evolocumab, a PCSK9 Inhibitor. Clin Pharmacokinet. 2018 Jul;57(7):769-779. doi: 10.1007/s40262-017-0620-7. PMID 29353350
- [Background] Sattar N, Toth PP, Blom DJ, Koren MJ, Soran H, Uhart M, Elliott M, Cyrille M, Somaratne R, Preiss D. Effect of the Proprotein Convertase Subtilisin/Kexin Type 9 Inhibitor Evolocumab on Glycemia, Body Weight, and New-Onset Diabetes Mellitus. Am J Cardiol. 2017 Nov 1;120(9):1521-1527. doi: 10.1016/j.amjcard.2017.07.047. Epub 2017 Jul 31. PMID 28844508
- [Background] Toth PP, Jones SR, Monsalvo ML, Elliott-Davey M, Lopez JAG, Banach M. Effect of Evolocumab on Non-High-Density Lipoprotein Cholesterol, Apolipoprotein B, and Lipoprotein(a): A Pooled Analysis of Phase 2 and Phase 3 Studies. J Am Heart Assoc. 2020 Mar 3;9(5):e014129. doi: 10.1161/JAHA.119.014129. Epub 2020 Mar 2. PMID 32114889
- [Background] Schludi B, Giugliano RP, Sabatine MS, Raal FJ, Teramoto T, Koren MJ, Stein EA, Wang H, Monsalvo ML. Time-averaged low-density lipoprotein cholesterol lowering with evolocumab: Pooled analysis of phase 2 trials. J Clin Lipidol. 2022 Jul-Aug;16(4):538-543. doi: 10.1016/j.jacl.2022.05.069. Epub 2022 Jun 6. PMID 35760720
- [Background] Hirayama A, Yamashita S, Ruzza A, Inomata H, Cyrille M, Lu C, Hamer AW, Yoshida M, Kiyosue A, Teramoto T. Long-Term Treatment With Evolocumab Among Japanese Patients - Final Report of the OSLER Open-Label Extension Studies. Circ J. 2019 Apr 25;83(5):971-977. doi: 10.1253/circj.CJ-19-0139. Epub 2019 Mar 29. PMID 30930429
- [Derived] Sabatine MS, Giugliano RP, Wiviott SD, Raal FJ, Blom DJ, Robinson J, Ballantyne CM, Somaratne R, Legg J, Wasserman SM, Scott R, Koren MJ, Stein EA; Open-Label Study of Long-Term Evaluation against LDL Cholesterol (OSLER) Investigators. Efficacy and safety of evolocumab in reducing lipids and cardiovascular events. N Engl J Med. 2015 Apr 16;372(16):1500-9. doi: 10.1056/NEJMoa1500858. Epub 2015 Mar 15. PMID 25773607
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This extension study was conducted at 188 centers in 18 countries. Participants were enrolled from one of five eligible phase 2 parent studies: 20101154 (NCT01375777), 20101155 (NCT01380730), 20090158 (NCT01375751), 20090159 (NCT01375764), and 20110231 (NCT01652703).
  Participants were enrolled from October 2011 to June 2013.
Pre-assignment Details: Participants were randomized in a 2:1 ratio, irrespective of their treatment assignments during the phase 2 parent study, to either evolocumab plus standard of care (SOC) or SOC alone. Randomization was stratified by the treatment to which the participant was randomized to in the parent study, ie evolocumab or control.
Groups:
- Standard of Care: Participants randomized to receive standard of care (SOC) treatment for the first year of the extension study (SOC-controlled period).
  At week 52 participants began treatment with evolocumab 420 mg QM for up to 4 years in the all-investigational product [all-IP] period.
- Evolocumab + SOC: Participants randomized to receive evolocumab 420 mg once a month plus standard of care for the first year of the extension study (SOC-controlled period).
  At week 52 participants continued treatment with evolocumab 420 mg QM for up to 4 years in the all-IP period.
Period: SOC-controlled Period (Year 1)
Arm/Group | Standard of Care | Evolocumab + SOC
Started | 442 | 882
Received Evolocumab | 0 | 881
Completed | 398 | 822
Not Completed | 44 | 60
Not completed — Withdrawal by Subject | 24 | 38
Not completed — Death | 2 | 1
Not completed — Sponsor Decision | 0 | 1
Not completed — Lost to Follow-up | 10 | 5
Not completed — Other | 8 | 13
Not completed — Reason Missing | 0 | 2
Period: All-IP Period (Years 2 to 5)
Arm/Group | Standard of Care | Evolocumab + SOC
Started | 398 | 822
Received Evolocumab | 374 | 777
Completed | 328 | 682
Not Completed | 70 | 140
Not completed — Lost to Follow-up | 21 | 30
Not completed — Withdrawal by Subject | 30 | 66
Not completed — Death | 3 | 13
Not completed — Sponsor Decision | 1 | 0
Not completed — Other | 14 | 31
Not completed — Reason Missing | 1 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set included all randomized participants
Groups:
- Standard of Care: Participants randomized to receive standard of care (SOC) treatment for the first year of the extension study (SOC-controlled period).
- Evolocumab + SOC: Participants randomized to receive evolocumab 420 mg once a month plus standard of care for the first year of the extension study (SOC-controlled period).
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Evolocumab + SOC | Total
Number analyzed (Participants) | 442 | 882 | 1324
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (11.5) | 56.9 (11.6) | 57.1 (11.6)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 307 | 632 | 939
  ≥ 65 years | 135 | 250 | 385
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 241 | 459 | 700
  Male | 201 | 423 | 624
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 39 | 52
  Not Hispanic or Latino | 429 | 843 | 1272
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 4
  Asian | 87 | 168 | 255
  Black or African American | 24 | 54 | 78
  Native Hawaiian or Other Pacific Islander | 2 | 5 | 7
  White | 325 | 648 | 973
  Other | 1 | 4 | 5
  Mixed Race | 0 | 2 | 2
Region [Count of Participants; unit: Participants]
  North America | 214 | 441 | 655
  Europe | 133 | 261 | 394
  Asia Pacific | 95 | 180 | 275
Parent Study Baseline Low-density Lipoprotein Cholesterol (LDL-C) Concentration [Mean (Standard Deviation); unit: mg/dL] | 144.6 (37.4) | 139.7 (36.7) | 141.3 (37.0)
Stratification Factor: Parent Study Treatment Assignment [Count of Participants; unit: Participants] — Randomization was stratified by the treatment to which a participant was randomized to in the parent study, according to the following:
  * randomized to evolocumab every 2 weeks (Q2W)
  * randomized to evolocumab QM
  * not randomized to evolocumab
  Participants
    Evolocumab once monthly (QM) | 193 | 387 | 580
    Evolocumab every 2 weeks (Q2M) | 129 | 256 | 385
    No evolocumab | 120 | 239 | 359

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Adverse event (AE) severity assessments were made using National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) grading, version 4.03, where grade 1 = mild AE, grade 2 = moderate AE, Grade 3 = severe AE, grade 4 = life-threatening AE and Grade 5 = death due to AE.
Time Frame: 52 weeks in the SOC-controlled period and up to 4 years in the All-IP period; actual median duration of treatment in the All-IP period was 46.9 months.
Population: All randomized participants (year 1) and randomized participants on study and who received at least 1 dose of evolocumab in the all-IP period (years 2-5).
Measure: Count of Participants; unit: Participants
Groups:
- SOC-controlled Period: Standard of Care: Participants randomized to receive standard of care (SOC) treatment for the first year of the extension study (SOC-controlled period).
- SOC-controlled Period: Evolocumab + SOC: Participants randomized to receive evolocumab 420 mg once a month plus standard of care for the first year of the extension study (SOC-controlled period).
- All-IP Period: SOC / Evolocumab + SOC: At week 52 participants began treatment with evolocumab 420 mg QM for up to 4 years during the all-IP period.
- All-IP Period: Evolocumab + SOC / Evolocumab + SOC: At week 52 participants continued treatment with evolocumab 420 mg QM for another 4 years during the all-IP period.
Arm/Group | SOC-controlled Period: Standard of Care | SOC-controlled Period: Evolocumab + SOC | All-IP Period: SOC / Evolocumab + SOC | All-IP Period: Evolocumab + SOC / Evolocumab + SOC
Number analyzed (Participants) | 442 | 882 | 374 | 777
Participants
  All adverse events | 327 | 728 | 342 | 718
  Adverse events ≥ grade 3 | 46 | 99 | 111 | 229
  Adverse events ≥ grade 4 | 2 | 11 | 8 | 28
  Serious adverse events | 30 | 72 | 76 | 172
  AEs leading to discontinuation of evolocumab | 0 | 28 | 16 | 27
  Fatal adverse events | 0 | 0 | 1 | 3

2. Secondary Outcome: Low-density Lipoprotein Cholesterol (LDL-C) Level at Week 24 and Week 52
Time Frame: Baseline of parent study and extension study weeks 24 and 52
Population: Participants randomized in study 20110110 and with available data at each time point.
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Control in Parent Study: SOC: Participants who received a control treatment in the parent study received standard of care treatment for the first year of the extension study.
- Control in Parent Study: Evolocumab + SOC: Participants who received a control treatment in the parent study received subcutaneous evolocumab 420 mg QM plus standard of care during the first year of the extension study.
- Evolocumab in Parent Study: SOC: Participants who received evolocumab in the parent study received standard of care treatment during the first year of the extension study.
- Evolocumab in Parent Study: Evolocumab + SOC: Participants who received evolocumab in the parent study received subcutaneous evolocumab 420 mg QM plus standard of care during the first year of the extension study.
Arm/Group | Standard of Care | Evolocumab + SOC | Control in Parent Study: SOC | Control in Parent Study: Evolocumab + SOC | Evolocumab in Parent Study: SOC | Evolocumab in Parent Study: Evolocumab + SOC
Number analyzed (Participants) | 442 | 882 | 120 | 239 | 322 | 643
mg/dL
  Parent Study Baseline | 144.6 (37.4) | 139.7 (36.7) | 147.7 (34.3) | 139.5 (33.6) | 143.4 (38.5) | 139.8 (37.8)
  Week 24: number analyzed (Participants) | 416 | 852 | 113 | 232 | 303 | 620
  Week 24 | 136.9 (41.5) | 64.1 (33.3) | 142.5 (44.7) | 63.9 (34.6) | 134.8 (40.2) | 64.2 (32.9)
  Week 52: number analyzed (Participants) | 399 | 826 | 113 | 224 | 286 | 602
  Week 52 | 140.5 (40.0) | 65.0 (34.4) | 143.1 (39.8) | 64.1 (33.2) | 139.4 (40.1) | 65.3 (34.9)

3. Secondary Outcome: Non-high-density Lipoprotein Cholesterol (Non-HDL-C) Level at Week 24 and Week 52
Time Frame: Baseline of parent study and extension study weeks 24 and 52
Population: Participants randomized in the extension study 20110110 and with available data at each time point.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Standard of Care | Evolocumab + SOC | Control in Parent Study: SOC | Control in Parent Study: Evolocumab + SOC | Evolocumab in Parent Study: SOC | Evolocumab in Parent Study: Evolocumab + SOC
Number analyzed (Participants) | 442 | 882 | 120 | 239 | 322 | 643
mg/dL
  Parent Study Baseline | 170.7 (43.0) | 165.1 (40.9) | 173.8 (39.6) | 165.5 (38.9) | 169.6 (44.2) | 165.0 (41.7)
  Week 24: number analyzed (Participants) | 416 | 852 | 113 | 232 | 303 | 620
  Week 24 | 161.4 (45.5) | 84.3 (37.7) | 166.9 (47.5) | 84.3 (39.0) | 159.4 (44.6) | 84.3 (37.3)
  Week 52: number analyzed (Participants) | 399 | 825 | 113 | 224 | 286 | 601
  Week 52 | 164.9 (44.5) | 85.3 (39.0) | 168.8 (45.3) | 85.0 (38.4) | 163.4 (44.1) | 85.4 (39.2)

4. Secondary Outcome: Apolipoprotein B Level at Week 24 and Week 52
Time Frame: Baseline of parent study and extension study weeks 24 and 52
Population: Participants randomized in the extension study 20110110 and with available data at each time point.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Standard of Care | Evolocumab + SOC | Control in Parent Study: SOC | Control in Parent Study: Evolocumab + SOC | Evolocumab in Parent Study: SOC | Evolocumab in Parent Study: Evolocumab + SOC
Number analyzed (Participants) | 442 | 882 | 120 | 239 | 322 | 643
mg/dL
  Parent Study Baseline | 113.2 (25.3) | 110.4 (23.8) | 115.4 (23.1) | 110.3 (22.4) | 112.4 (26.0) | 110.4 (24.3)
  Week 24: number analyzed (Participants) | 416 | 852 | 113 | 232 | 303 | 620
  Week 24 | 107.9 (26.3) | 60.8 (23.3) | 110.5 (27.0) | 60.7 (23.9) | 106.9 (26.0) | 60.9 (23.1)
  Week 52: number analyzed (Participants) | 401 | 834 | 113 | 227 | 288 | 607
  Week 52 | 109.5 (26.8) | 61.6 (23.5) | 110.7 (26.3) | 61.7 (23.0) | 109.1 (27.0) | 61.6 (23.7)

5. Secondary Outcome: Total Cholesterol/HDL-C Ratio at Week 24 and Week 52
Time Frame: Baseline of parent study and extension study weeks 24 and 52
Population: Participants randomized in the extension study 20110110 and with available data at each time point.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Standard of Care | Evolocumab + SOC | Control in Parent Study: SOC | Control in Parent Study: Evolocumab + SOC | Evolocumab in Parent Study: SOC | Evolocumab in Parent Study: Evolocumab + SOC
Number analyzed (Participants) | 442 | 882 | 120 | 239 | 322 | 643
ratio
  Parent Study Baseline | 4.516 (1.617) | 4.386 (1.393) | 4.458 (1.345) | 4.388 (1.340) | 4.538 (1.708) | 4.386 (1.413)
  Week 24: number analyzed (Participants) | 416 | 852 | 113 | 232 | 303 | 620
  Week 24 | 4.198 (1.536) | 2.603 (0.978) | 4.192 (1.408) | 2.594 (0.970) | 4.201 (1.584) | 2.607 (0.982)
  Week 52: number analyzed (Participants) | 399 | 825 | 113 | 224 | 286 | 601
  Week 52 | 4.277 (1.652) | 2.626 (1.025) | 4.252 (1.434) | 2.622 (1.033) | 4.286 (1.733) | 2.628 (1.023)

6. Secondary Outcome: Apolipoprotein B/Apolipoprotein A1 Ratio at Week 24 and Week 52
Time Frame: Baseline of parent study and extension study weeks 24 and 52
Population: Participants randomized in the extension study 20110110 and with available data at each time point.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Standard of Care | Evolocumab + SOC | Control in Parent Study: SOC | Control in Parent Study: Evolocumab + SOC | Evolocumab in Parent Study: SOC | Evolocumab in Parent Study: Evolocumab + SOC
Number analyzed (Participants) | 442 | 882 | 120 | 239 | 322 | 643
ratio
  Parent Study Baseline | 0.759 (0.237) | 0.739 (0.217) | 0.764 (0.201) | 0.735 (0.212) | 0.757 (0.249) | 0.741 (0.218)
  Week 24: number analyzed (Participants) | 416 | 852 | 113 | 232 | 303 | 620
  Week 24 | 0.717 (0.242) | 0.386 (0.178) | 0.715 (0.222) | 0.385 (0.183) | 0.718 (0.250) | 0.387 (0.176)
  Week 52: number analyzed (Participants) | 401 | 834 | 113 | 227 | 288 | 607
  Week 52 | 0.726 (0.256) | 0.394 (0.185) | 0.719 (0.216) | 0.393 (0.186) | 0.729 (0.271) | 0.394 (0.185)

ADVERSE EVENTS:
Time Frame: 52 weeks in the SOC-controlled period and up to 4 years in the All-IP period; median duration of treatment in the All-IP period was 46.9 months.
Description: Adverse events are reported for all randomized participants in the SOC-controlled period (year 1) and for all participants who entered the All-IP period (years 2-5).
  Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- SOC-controlled Period: SOC: Participants received standard of care (SOC) treatment for the first year of the study (SOC-controlled period).
- SOC-controlled Period: Evolocumab + SOC: Participants received evolocumab 420 mg once a month for the first year of the study (SOC-controlled period).
- All-IP Period: SOC / Evolocumab: At week 52 participants began treatment with evolocumab 420 mg QM for up to 4 years during the all-IP period.
- All-IP Period: Evolocumab + SOC / Evolocumab: At week 52 participants continued treatment with evolocumab 420 mg QM for another 4 years during the all-IP period.
- All-IP Period: Total: All participants in the All-IP period who received evolocumab 420 mg QM for up to 4 years.
Arm/Group | SOC-controlled Period: SOC | SOC-controlled Period: Evolocumab + SOC | All-IP Period: SOC / Evolocumab | All-IP Period: Evolocumab + SOC / Evolocumab | All-IP Period: Total
All-Cause Mortality (participants affected / at risk) | 2/442 | 1/882 | 3/398 | 13/822 | 16/1220
Serious Adverse Events (participants affected / at risk) | 30/442 | 72/882 | 78/398 | 181/822 | 259/1220
Other Adverse Events (participants affected / at risk) | 217/442 | 513/882 | 311/398 | 626/822 | 937/1220
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOC-controlled Period: SOC (N=442) | SOC-controlled Period: Evolocumab + SOC (N=882) | All-IP Period: SOC / Evolocumab (N=398) | All-IP Period: Evolocumab + SOC / Evolocumab (N=822) | All-IP Period: Total (N=1220)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Angina pectoris (Cardiac disorders) | 2 | 4 | 1 | 9 | 10
Angina unstable (Cardiac disorders) | 0 | 1 | 1 | 1 | 2
Aortic valve disease (Cardiac disorders) | 0 | 0 | 0 | 2 | 2
Aortic valve disease mixed (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Aortic valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Aortic valve sclerosis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Aortic valve stenosis (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 2 | 7 | 9
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 1 | 1
Atrial thrombosis (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 1 | 2
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 2 | 2
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 1 | 2
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1 | 2 | 4 | 6
Coronary artery embolism (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 1 | 1 | 2 | 3
Mitral valve disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Mitral valve disease mixed (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 2 | 2
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Nodal rhythm (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Thyroid mass (Endocrine disorders) | 1 | 0 | 0 | 0 | 0
Thyroiditis acute (Endocrine disorders) | 0 | 0 | 0 | 1 | 1
Cataract (Eye disorders) | 0 | 0 | 2 | 2 | 4
Cataract cortical (Eye disorders) | 0 | 1 | 0 | 0 | 0
Corneal defect (Eye disorders) | 0 | 0 | 0 | 1 | 1
Eyelid ptosis (Eye disorders) | 0 | 0 | 0 | 1 | 1
Keratitis (Eye disorders) | 1 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Brunner's gland hyperplasia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 2
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 2
Ileus paralytic (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 2
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 3
Lumbar hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Obstructive pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Oesophageal spasm (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 2
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Splenic artery aneurysm (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Tooth impacted (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 4 | 1 | 6 | 7
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 1
Hypothermia (General disorders) | 0 | 0 | 1 | 0 | 1
Mass (General disorders) | 0 | 0 | 0 | 1 | 1
Nodule (General disorders) | 0 | 0 | 1 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 4 | 0 | 7 | 7
Organ failure (General disorders) | 0 | 0 | 0 | 1 | 1
Pain (General disorders) | 0 | 0 | 0 | 1 | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1
Biliary dyskinesia (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 2 | 1 | 3
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 4 | 4
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 4 | 5
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 2
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1
Contrast media allergy (Immune system disorders) | 0 | 1 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 1
Abscess limb (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Appendiceal abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Appendicitis (Infections and infestations) | 1 | 5 | 2 | 3 | 5
Arthritis bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Arthritis infective (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Bacterial pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 2 | 2 | 4
Bursitis infective (Infections and infestations) | 0 | 0 | 0 | 2 | 2
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 2 | 2
Cellulitis staphylococcal (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Chronic sinusitis (Infections and infestations) | 0 | 1 | 1 | 0 | 1
Clostridial infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Cystitis (Infections and infestations) | 1 | 0 | 0 | 1 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 1 | 2
Endocarditis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Escherichia sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 2 | 2
Gastroenteritis bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Groin abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Infective spondylitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Joint abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Meningitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Ophthalmic herpes simplex (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 3 | 2 | 4 | 6
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Pyelonephritis (Infections and infestations) | 0 | 1 | 1 | 3 | 4
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Rocky mountain spotted fever (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Streptococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 4 | 4
Anaesthetic complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 2
Cardiac contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 2 | 4
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 2
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Intervertebral disc injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1 | 2
Procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Procedural nausea (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Procedural vomiting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Pulmonary contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 1 | 3
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Tendon injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Urinary retention postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 3 | 4
Electrocardiogram ST segment abnormal (Investigations) | 0 | 1 | 0 | 0 | 0
HIV test positive (Investigations) | 0 | 0 | 0 | 1 | 1
Heart rate increased (Investigations) | 0 | 0 | 1 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 0 | 1 | 1 | 2
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1 | 1
Weight decreased (Investigations) | 0 | 0 | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 3 | 2 | 0 | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 3 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 3 | 4
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 2
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 1 | 3
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 3 | 5 | 9 | 14
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 2
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 3 | 4
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 1 | 3
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 5 | 6
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2 | 1 | 3
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 1
Hairy cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Intraductal papilloma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 2 | 2
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 2 | 2
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Mantle cell lymphoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2 | 2
Myxoid liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2 | 2
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2 | 4 | 6
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 2
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 1
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Brain stem haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Cerebral thrombosis (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Cervical radiculopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 2 | 0 | 2
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Facial paralysis (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Guillain-Barre syndrome (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Lumbar radiculopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Motor neurone disease (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Myelopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Presyncope (Nervous system disorders) | 0 | 2 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Spinal claudication (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Syncope (Nervous system disorders) | 0 | 2 | 0 | 4 | 4
Tension headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Trigeminal neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0
Alcohol abuse (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1
Depression (Psychiatric disorders) | 0 | 1 | 1 | 1 | 2
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 0 | 2 | 2
Bladder prolapse (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1
Calculus bladder (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 2
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 1 | 3 | 4
Renal artery stenosis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 2 | 0 | 1 | 1
Cystocele (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 1
Uterine prolapse (Reproductive system and breast disorders) | 1 | 0 | 1 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 4 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 2
Laryngeal polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 4 | 5
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1
Cholecystectomy (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 1
Knee arthroplasty (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 1
Medical device removal (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 1
Accelerated hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Aortic aneurysm (Vascular disorders) | 0 | 0 | 1 | 0 | 1
Aortic stenosis (Vascular disorders) | 0 | 1 | 1 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 2 | 2
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 1
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 1 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 0 | 1 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 0 | 1 | 1
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SOC-controlled Period: SOC (N=442) | SOC-controlled Period: Evolocumab + SOC (N=882) | All-IP Period: SOC / Evolocumab (N=398) | All-IP Period: Evolocumab + SOC / Evolocumab (N=822) | All-IP Period: Total (N=1220)
Diarrhoea (Gastrointestinal disorders) | 11 | 41 | 33 | 61 | 94
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 13 | 23 | 20 | 32 | 52
Nausea (Gastrointestinal disorders) | 4 | 23 | 23 | 32 | 55
Fatigue (General disorders) | 5 | 31 | 16 | 43 | 59
Bronchitis (Infections and infestations) | 17 | 48 | 40 | 94 | 134
Cystitis (Infections and infestations) | 9 | 15 | 25 | 39 | 64
Influenza (Infections and infestations) | 24 | 57 | 47 | 81 | 128
Nasopharyngitis (Infections and infestations) | 64 | 148 | 122 | 236 | 358
Sinusitis (Infections and infestations) | 15 | 32 | 31 | 68 | 99
Upper respiratory tract infection (Infections and infestations) | 29 | 72 | 57 | 118 | 175
Contusion (Injury, poisoning and procedural complications) | 10 | 15 | 25 | 35 | 60
Procedural pain (Injury, poisoning and procedural complications) | 4 | 4 | 20 | 23 | 43
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 | 59 | 63 | 109 | 172
Back pain (Musculoskeletal and connective tissue disorders) | 22 | 62 | 51 | 117 | 168
Muscle spasms (Musculoskeletal and connective tissue disorders) | 10 | 25 | 21 | 39 | 60
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 12 | 28 | 19 | 62 | 81
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 22 | 27 | 54 | 81
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 | 44 | 32 | 70 | 102
Dizziness (Nervous system disorders) | 12 | 18 | 20 | 51 | 71
Headache (Nervous system disorders) | 12 | 54 | 28 | 44 | 72
Cough (Respiratory, thoracic and mediastinal disorders) | 19 | 41 | 40 | 77 | 117
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 | 24 | 14 | 42 | 56
Hypertension (Vascular disorders) | 20 | 52 | 40 | 99 | 139

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2015-11-12): https://cdn.clinicaltrials.gov/large-docs/80/NCT01439880/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-22): https://cdn.clinicaltrials.gov/large-docs/80/NCT01439880/SAP_001.pdf